CLINICAL TRIAL: NCT02967042
Title: Chronic Kidney Disease and Bone - Correlation Between 18F-PET-TT Imaging and Histomorphometry of Bone in Patients With Chronic Kidney Disease and Secondary Hyperparathyroidism
Brief Title: Chronic Kidney Disease and Bone - Correlation Between 18F-PET-TT Imaging and Histomorphometry of Bone in CKD Patients
Acronym: CKD-Bone
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: T239/2016
Record Dates: First submitted 2016-09-22; First posted 2016-11-17 (Estimated); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 18F-PET-TT (Other)
  Interventions: Device: 18F-PET-TT

INTERVENTIONS:
Device: 18F-PET-TT — can 18F-PET-TT be used as an diagnostic tool in patients with CKD-MBD

SUMMARY:
Chronic kidney disease (CKD) is an increasing public health problem and the number of patient with chronic kidney disease is increasing worldwide. Bone abnormalities are found almost universally in patients with CKD requiring dialysis and in the majority of patients with CKD stages 3-5. Chronic kidney disease-mineral bone disorder (CKD-MBD) is a complex disorder of bone and mineral metabolism, which is associated with disorder in circulating levels of hormones and development of secondary hyperparathyroid disease. The abnormalities of mineral homeostasis impair bone remodeling and mineralization and results in cortical and trabecular defects and an increased fracture risk. There is also an association with increased morbidity and mortality. CKD-MBD is also associated with development of calcification of the blood vessels. During the last decade it has been increasingly acknowledged that mineral and bone disorder contribute to the excessively high cardiovascular morbidity and mortality in patients with chronic kidney disease.

The diagnosis of mineral bone disorder and the underlying bone histology in CKD patients is challenging. The treatment of renal osteodystrophy (ROD) and especially the treatment of fractures in this patient group, depends on the underlying bone histopathology and bone turnover. The gold standard for diagnosing the subtypes of ROD is bone biopsy, but it is invasive and requires considerable expertise regarding quantitative histomorphometry and interpretation. Plasma parathormone (PTH) measurement is commonly used to evaluate these patients, and generally extremely high or low PTH levels predict the underlying bone disorder. Still PTHs ability to correctly estimate turnover in bone is limited. Several biomarkers such as tartrate-resistant acid phosphatase 5b (TRAP5b) and procollagen type 1 N-terminal propetide (PINP) has been investigated, but no biomarker in clinical use has yet been proven suitable or superior to PTH to estimate overall bone histology.

18F-NaF positron emission tomography (18F-NaF PET) is a noninvasive quantitative imaging technique that allows assessment of regional bone turnover at clinically relevant sites. 18F-NaF is a bone-seeking tracer, which reflects remodeling of bone and osteoblast activity25. 18F-NaF serves as an efficient tracer to measure metabolic changes in bone. A correlation between histomorphometric markers such as bone formation rate (BFR) and tracer activity in the 18F- NaF PET scan in CKD patients has previously been shown in one small study.

This study's goal is to evaluate, if 18-NaF-Positron emission tomography-computed tomography (18F-PET-TT) can be used in the assessment of CKD patients. The hypothesis is that 18F-PET-TT correlates with the histomorphometry of bone biopsy and with the calcification score in CKD patients and that 18F-PET-TT maybe can be used as a diagnostic imaging technique in the future.

DETAILED DESCRIPTION:
This is a cross-sectional prospective study. 10 - 20 patients with secondary/tertiary hyprparathyreoidism on oeritoneal dialysis, hemodialysis, predialysis patients and patients, who have received a kidney transplant will be included,. Data collection in the dialysis group is finnished and the first article published (Aaltonen et al, Bone 2020). A control group was recruited for validation of the PET-method.

All participants undergo a 18F-PET-TT scan. PET, with the short half-life bone seeking 18F-Sodium Fluoride (18F-NaF), provide an unique way of assessment of regional bone metabolism. 18F-NaF binds to sights of new bone formation and serves as a marker of bone blood flow and osteoblastic activity. A dynamic 18F-PET-TT imaging is first done of the lumbar region of the spine, following with a static PET-TT and also measurement of calcification score using PET-TT. 18F-NaF is injected intravenously by direct venipuncture or intravenous catheter. All the patients are also asked for permission to use DNA-samples if needed.

Blood tests measuring the bone formation and turnover will be taken during the normal clinical controls of the patients or at the latest wheb the bone biopsy is takekn. Echocardiogram, which is reasonable sensitive, is done to detect and evaluate valvular calcification. Bone biopsy is done in the day care unit within one month from the PET-scan. To obtain information about dynamic parameters of the bone, the patients had double labeling with tetracycline. The biopsy is taken in local anesthesia from the anterior iliac spine vertically.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severely decreased kidney function (eGRF below 20ml/min) with secondary hyperparathyroidism. In addition a group of healthy volunteers.

Exclusion Criteria:

* Pregnancy, parathyroidectomy, biphosphonate-medication.

Ages: 25 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-12-17 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Evidence of kidney patients adynamic or hyperdynamic bone disease assessed by 18F-PET-TT | 3 years
  18F-PET correlates with histomorphometric markers in bone biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Kaj Metsärinne, LT, Study Director — Senior physician /TYKS - nefrologia ja dialyysihoidot
Locations (1):
- TYKS/nefrologia ja dialyysihoidot, Turku, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aaltonen L, Koivuviita N, Seppanen M, Kroger H, Tong X, Loyttyniemi E, Metsarinne K. Association between bone mineral metabolism and vascular calcification in end-stage renal disease. BMC Nephrol. 2022 Jan 3;23(1):12. doi: 10.1186/s12882-021-02652-z. PMID 34979983
- See also: Correlation between 18F-Sodium Fluoride positron emission tomography and bone histomorphometry in dialysis patients — https://doi.org/10.1016/j.bone.2020.115267